CLINICAL TRIAL: NCT05911555
Title: A Single-Center Pilot Study To Evaluate the Effects of a Challenge Model on Mucin 16 Levels in Dry Eye Subjects Compared to Normal Subjects
Brief Title: Mucin Levels in Dry Eye and Normal Populations
Status: Completed | Type: Observational
Sponsor: ORA, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-270-0004
Record Dates: First submitted 2013-07-30; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tear collection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-Dry Eye Subjects: Subjects with no reported history of dry eye disease will be enrolled
- Dry Eye Disease: Subjects who have been diagnosed with dry eye disease in a previous trial will be enrolled.

SUMMARY:
The purpose of this study is to evaluate changes in ocular mucin levels in response to a drying environment in subjects with dry eye disease as well as patients who report no history of dry eye disease.

It is expected that exposure to the dry environment will alter mucin levels in different ways when comparing the two groups.

DETAILED DESCRIPTION:
This is a single-center, two visit, pilot, drying environment study (CAE). There will be two different groups of subjects enrolled into this study: dry eye subjects and subjects with no prior diagnosis of dry eye.

All subjects will undergo safety and dry eye assessments as well as tear collection prior to and after being exposed to a dry environment. They will also return the following day to undergo dry eye assessments, tear collection, and safety procedures again.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female of any race, at least 18 years of age at Visit 1.
* Have provided verbal and written informed consent.
* Have a best corrected visual acuity of +0.70 logMAR or better in both eyes at Visit 1, as assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) chart.
* If a woman of childbearing potential, have a negative urine pregnancy test at Visit 1 and agree to use a medically acceptable form of birth control throughout the study duration . [Females are considered of childbearing potential unless they are surgically sterilized (bilateral tubal ligation, hysterectomy or bilateral oophorectomy) or post-menopausal (at least 12 months since last menses).]
* Have previously completed a recent trial OR not completed a recent trial AND report no symptoms of dry eye disease.

Exclusion Criteria:

* Have planned surgery during trial period
* Female currently pregnant, planning a pregnancy or lactating
* Use of disallowed medications
* Have ocular infections, or ocular conditions that could affect study parameters
* Have used an investigational drug or device within 30 days of start of study
* Female that is currently pregnant, planning a pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with dry eye will be selected from a previous trial and subjects without dry eye will be also be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2013-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Mucin levels assayed from collected tears | 10-30 minutes Post CAE at Visit 1
  Tears will be collected and mucin will be measured after subjects are exposed to the CAE.
Mucin levels assayed from collected tears | 24 hours after being exposed to the CAE
  Tears will be collected and mucin will be measured 24 hours after being exposed to the CAE.

SECONDARY OUTCOMES:
Fluorescein staining | pre-CAE
  staining will be measured to detect presence of Superficial Punctate Keratitis and Confluency using Ora Calibra™ Corneal and Conjunctival Staining Scales
Fluorescein staining | 10-30 minutes Post CAE
  Staining will be measured to detect presence of Superficial Punctate Keratitis and Confluency using Ora Calibra™ Corneal and Conjunctival Staining Scales
Fluorescein staining | 24 hours post-CAE
  Staining will be measured measured to detect presence of Superficial Punctate Keratitis and Confluency using Ora Calibra™ Corneal and Conjunctival Staining Scales
Lissamine staining | pre-CAE
  Staining will be measured to detect presence of Superficial Punctate Keratitis and Confluency using Ora Calibra™ Corneal and Conjunctival Staining Scales
Lissamine staining | 10-30 minutes Post CAE
  Staining will be measured to detect presence of Superficial Punctate Keratitis and Confluency using Ora Calibra™ Corneal and Conjunctival Staining Scales
Lissamine staining | 24 hours post-CAE
  Staining will be measured to detect presence of Superficial Punctate Keratitis and Confluency using Ora Calibra™ Corneal and Conjunctival Staining Scales
Presence of conjunctival redness | pre-CAE
  conjunctival redness will be assessed by Ora Calibra™ Conjunctival Redness Scale
Presence of conjunctival redness | 10-30 minutes Post CAE
  conjunctival redness will be assessed by Ora Calibra™ Conjunctival Redness Scale
Presence of conjunctival redness | 24 hours post-CAE
  conjunctival redness will be assessed by Ora Calibra™ Conjunctival Redness Scale
Tear Film Break Up Time | pre-CAE
  Tear Film Break Up Time
Tear Film Break Up Time | 10-30 minutes Post CAE
  Tear Film Break Up Time
Tear Film Break Up Time | 24 hours post-CAE
  Tear Film Break Up Time
Blink Rate Analysis | pre-CAE
  Blink Rate Analysis
Blink Rate Analysis | 10-30 minutes Post CAE
  Blink Rate Analysis
Blink Rate Analysis | 24 hours post-CAE
  Blink Rate Analysis
Symptom Collection | pre-CAE
  Symptom Collection
Symptom Collection | 10-30 minutes Post CAE
  Symptom Collection
Symptom Collection | 24 hours post-CAE
  Symptom Collection
Ora Calibra Ocular Protection Index 2.0 | pre-CAE
  Ora Calibra Ocular Protection Index 2.0
Ora Calibra Ocular Protection Index 2.0 | 10-30 minutes Post CAE
  Ora Calibra Ocular Protection Index 2.0
Ora Calibra Ocular Protection Index 2.0 | 24 hours post-CAE
  Ora Calibra Ocular Protection Index 2.0
Schirmer's Test | End of Visit 2 (Day 1 of study)
  Schirmer's Test

OTHER OUTCOMES:
Adverse Event Query | Beginning of Visit 1 (Day 0)
  All adverse events that are reported during these visits will be followed up on until they are resolved or stabilized
Adverse Event Query | End of Visit 2 (Day 1)
  All adverse events that are reported during these visits will be followed up on until they are resolved or stabilized
Best Corrected Visual Acuity | Beginning and end of Visit 1 (Day 0)
  Best Corrected Visual Acuity
Best Corrected Visual Acuity | Beginning of Visit 2 (Day 1)
  Best Corrected Visual Acuity
Urine Pregnancy test | Beginning of Visit 1 (Day 0)
  Urine Pregnancy test

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States